CLINICAL TRIAL: NCT02528656
Title: Physiological Assessments During Non Operative Treatment on the Chest Wall Deformities. Pectus Excavatum Pectus-Carinatum. Single-center Study
Brief Title: Physiological Assessments During Non Operative Treatment on the Chest Wall Deformities
Acronym: PECTUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: MEDICALEX (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1408081; 2014-A00841-46 (Other: ANSM)
Record Dates: First submitted 2015-08-13; First posted 2015-08-19 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pectus Excavatum; Pectus Carinatum
Keywords: Pectus Excavatum; Pectus Carinatum; Vacuum Bell; Dynamic compression system; Hearth variability; Autonomic Nervous System
MeSH Terms: conditions — Funnel Chest; Pectus Carinatum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pectus Excavatum (Experimental): Patients with pectus excavatum who do not require surgery, will be treated with the Vacuum bell device.
  Interventions: Device: Vacuum Bell
- Pectus Carinatum (Experimental): Patients with pectus carinatum who do not require surgery, will be treated with the Dynamic Compression System.
  Interventions: Device: Dynamic Compression System

INTERVENTIONS:
Device: Vacuum Bell — Patients will be submitted to a negative pressure treatment with the Vacuum Bell device.
  Arms: Pectus Excavatum
Device: Dynamic Compression System — Patients will be submitted to a dynamic compression system.
  Arms: Pectus Carinatum

SUMMARY:
The physiological assessment in non-operative treatment on chest wall deformities, are still unclear today. These functional benefits outweigh the aesthetic benefits associated with anatomical improvement. The functional benefits, ventilation, hemodynamic and neurologic, have never been evaluated.

Assessment of Effects on parasympathetic activity of the autonomic nervous system, global health criterion measured by noninvasive methods.

Anatomic evaluation, between the initial and final assessment by objective measures 1) of the chest wall by MRI, and 2) of the heart by echocardiography.

Noninvasive physiological assessment at rest and during exercise in respiratory function exploration flows and volumes, cardiac function by flow measurement, and overall metabolic function test effort (VO2max). Subjective assessment of functional gain between the initial and final balance sheet, based on EVA scales, valued by patients, parents and doctors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pectus excavatum or pectus carinatum who does not require surgery
* Patient with sufficient displacement of the chest wall during an initial test carried out during the first consultation :For pectus carinatum correction must be obtained with a pressure lower than 9 psi (pound per square inch). For pectus excavatum less than 250 mbar depression.
* Signed informed consent
* Subject (or parents) affiliated to the French National Health Insurance

Exclusion Criteria:

* Skeletal disease, disturbing bone strength as osteogenesis imperfect and osteoporosis.
* Uncontrolled coagulopathies.
* Marfan syndrome, with mitral valve prolapse for pectus Excavatum.
* Atrial fibrillation
* Taking antiarrhythmic drug.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-01-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
High frequency normalized index (HFnu) | One month after the end of treatment
  It is a reflect of the RR short term heart rate variability (HRV) in the frequency domain. It is measured with a ECG Holter monitor

SECONDARY OUTCOMES:
Low frequency (LF and LFnu) | One month after the end of treatment
  It is another index of RR heart rate variability (HRV) measured with a ECG Holter monitor.
LF/HF ratio | One month after the end of treatment
  It is another index of RR heart rate variability (HRV) measured with a ECG holter monitor.
Blood pressure - Baroreflex | One month after the end of treatment
  Measure of autonomic function (parasympathetic activity) - quantified via changes in blood pressure
Lung residual volume | One month after the end of treatment
  It is expressed in litres and is measured with a plethysmograph during a pulmonary function testing.
Maximum flow | One month after the end of treatment
  It is expressed in litres per minute and is measured during a pulmonary function testing. The patient is seated and his/her nose is blocked with a clamp. He/She must blow as fast and as hard as possible.
Aerobic maximum power | One month after the end of treatment
  It is measured by a stress test (incremental exercise)
Maximum heart rate | One month after the end of treatment
  It is measured by a stress test (incremental exercise)
Left ventricular ejection fraction | One month after the end of treatment
  It is measured by an echocardiography
Severity index of the anatomical damage | One month after the end of treatment
  It is measured by a thoracic MRI. It is the ratio between the thoracic width and the distance sternum/spine.
Nuss Questionnaire | One month after the end of treatment
  It is a depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Manuel LOPEZ, MD, Study Chair — CHU de SAINT-ETIENNE; Arnaud PATOIR, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No